CLINICAL TRIAL: NCT01491607
Title: Immunogenicity and Safety Study of a Three-Dose BioThrax® Regimen for Post-Exposure Prophylaxis in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBS.AVA.006; HHSO100200700037C (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Anthrax
Keywords: post-exposure prophylaxis; toxin neutralization assay
MeSH Terms: conditions — Anthrax | interventions — Biothrax; Anthrax Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioThrax (0.5 mL, on days 0, 14, and 28) (Experimental)
  Interventions: Biological: BioThrax

INTERVENTIONS:
Biological: BioThrax — BioThrax, 0.5 mL administered subcutaneously on days 0, 14, and 28.
  Other Names: Anthrax Vaccine Adsorbed (AVA)

SUMMARY:
The purpose of this Phase 3 clinical trial is to evaluate the immunogenicity and safety of BioThrax anthrax vaccine in healthy adults following 3 doses of BioThrax. Results of this study will be used to support a post-exposure prophylaxis (PEP) indication for BioThrax.

This study will be conducted in the United States (U.S.), in 200 healthy male and female volunteer subjects ages 18 to 65 years.

The duration of study participation for each individual subject will be approximately 128 days (4.25 months), including a screening period of approximately 28 days followed by 100 days on study.

DETAILED DESCRIPTION:
BioThrax® (also called Anthrax Vaccine Adsorbed or AVA) is the only FDA-licensed vaccine for the prevention of anthrax infection. This study will evaluate the immunogenicity of the vaccine using a post-exposure vaccination schedule. Correlations will be drawn to immunogenicity and survival data from animal models to demonstrate that BioThrax® can elicit a protective immune response for PEP.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years of age, inclusive, at the time of enrollment.
* Be in good health as determined by the investigator from medical history and a physical examination.
* If a pre-menopausal female, must be using acceptable methods of birth control.
* Have all hematology and chemistry parameters (measured at Screening) within the laboratory's normal range.
* Be willing and able to return for all visits and blood collections for the duration of the study.
* Have read, understood and signed an informed consent form.

Exclusion Criteria:

* Prior immunization with anthrax vaccine or known exposure to anthrax organisms.
* Intend to enlist in the military during the study.
* Have a known allergy to aluminum hydroxide, formaldehyde, benzethonium chloride, or latex.
* Plan to receive experimental products at any time during the study.
* Have received a live vaccine in the 30 days before study entry.
* Plan to receive a live vaccine at any time during the study.
* Have ongoing drug abuse/dependence (including alcohol) issues and/or test positive in a urine drug screen for amphetamines, barbiturates, cocaine or opiates;
* Have received immunosuppressive therapy (including systemic steroids) within 3 months prior to study entry.
* Have a condition known to produce or be associated with immunosuppression.
* Have received cytotoxic therapy in the previous 5 years.
* A medical condition that, in the opinion of the Principal Investigator (PI), could adversely impact the subject's participation, safety, or conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hopkins, MD, MPH, TM, Principal Investigator — Emergent BioSolutions Inc.
Locations (4):
- United States (4):
  - Miami Research Associates, Miami, Florida
  - Rochester Clinical Research, Rochester, New York
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 9 November 2011 to 9 May 2012 at four medical centers in the U.S.
Pre-assignment Details: All enrolled participants met the inclusion and exclusion criteria.
Groups:
- BioThrax: Participants 18 to 65 years of age who received at least one dose of BioThrax (0.5 mL) subcutaneously (SC).
Period: Overall Study
Arm/Group | BioThrax
Started | 200
Completed | 190
Not Completed | 10
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Participants 18 to 65 years of age who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
Groups:
- BioThrax - Site 01: Subjects from Site 01 who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
- BioThrax - Site 02: Subjects from Site 02 who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
- BioThrax - Site 03: Subjects from Site 03 who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
- BioThrax - Site 04: Subjects from Site 04 who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
- Total: Total of all reporting groups
Arm/Group | BioThrax - Site 01 | BioThrax - Site 02 | BioThrax - Site 03 | BioThrax - Site 04 | Total
Number analyzed (Participants) | 45 | 34 | 56 | 49 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 1 | 3
  Between 18 and 65 years | 44 | 33 | 56 | 48 | 181
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (11.41) | 36.7 (10.97) | 32.7 (9.89) | 34.2 (11.09) | 33.7 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 29 | 22 | 92
  Male | 23 | 15 | 27 | 27 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 15 | 1 | 2 | 20
  Not Hispanic or Latino | 43 | 19 | 55 | 47 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 20 | 49 | 45 | 156
  Black or African American | 0 | 14 | 3 | 3 | 20
  Asian | 2 | 0 | 2 | 1 | 5
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 45 | 34 | 56 | 49 | 184

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a TNA Response of a Predefined Threshold Value at Day 63 (5 Weeks Following the Third Vaccination on Day 28).
Description: Neutralizing antibody levels in blinded serum samples were measured using a validated anthrax lethal toxin neutralization assay. The primary assay endpoint was the 50% neutralization factor (TNA NF50), which is calculated as the ratio of the 50% effective dose (ED50) of the test sample to the ED50 of a reference serum.
Time Frame: Day 63 +/- 2 days
Population: Subjects who received all three doses of BioThrax within the allowable time window and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by Sponsor) on Day 63 were excluded.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- BioThrax: Participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
- BioThrax - Male: Male participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population..
- BioThrax - Female: Female participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population..
- BioThrax - ≤ 30 Years of Age: Participants ≤ 30 Years of Age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population..
- BioThrax- > 30 Years of Age: Participants > 30 Years of Age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
- BioThrax - Caucasian: Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population..
- BioThrax - Non-Caucasian: Non-Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population..
- BioThrax - Site 01: Participants enrolled at Site 01 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
- BioThrax - Site 02: Participants enrolled at Site 02 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
- BioThrax - Site 03: Participants enrolled at Site 03 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
- BioThrax - Site 04: Participants enrolled at Site 04 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 63 were excluded from the Primary Per-Protocol Population.
Arm/Group | BioThrax | BioThrax - Male | BioThrax - Female | BioThrax - ≤ 30 Years of Age | BioThrax- > 30 Years of Age | BioThrax - Caucasian | BioThrax - Non-Caucasian | BioThrax - Site 01 | BioThrax - Site 02 | BioThrax - Site 03 | BioThrax - Site 04
Number analyzed (Participants) | 184 | 92 | 92 | 90 | 94 | 156 | 28 | 45 | 34 | 56 | 49
percentage of participants | 71.2 [64.1 to 77.6] | 68.5 [58.0 to 77.8] | 73.9 [63.7 to 82.5] | 76.7 [66.6 to 84.9] | 66.0 [55.5 to 75.4] | 73.7 [66.1 to 80.4] | 57.1 [37.2 to 75.5] | 91.1 [78.8 to 97.5] | 67.6 [49.5 to 82.6] | 69.6 [55.9 to 81.2] | 57.1 [42.2 to 71.2]

2. Secondary Outcome: Percentage of Subjects Achieving a TNA Response of a Predefined Threshold Value at Day 70.
Description: as for outcome 1
Time Frame: Day 70 +/- 2 days
Population: Participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- BioThrax - Day 70: Participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Male: Male participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Female: Female participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - ≤ 30 Years of Age: Participants ≤ 30 Years in age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - > 30 Years of Age: Participants > 30 Years in age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Caucasian: Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Non-Caucasian: Non-Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Site 01: Participants enrolled at Site 01, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Site 02: Participants enrolled at Site 02, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Site 03: Participants enrolled at Site 03, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
- BioThrax - Site 04: Participants enrolled at Site 04, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 70 ± 2 days. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Day 70 were excluded.
Arm/Group | BioThrax - Day 70 | BioThrax - Male | BioThrax - Female | BioThrax - ≤ 30 Years of Age | BioThrax - > 30 Years of Age | BioThrax - Caucasian | BioThrax - Non-Caucasian | BioThrax - Site 01 | BioThrax - Site 02 | BioThrax - Site 03 | BioThrax - Site 04
Number analyzed (Participants) | 183 | 90 | 93 | 88 | 95 | 156 | 27 | 43 | 33 | 57 | 50
percentage of participants | 57.9 [50.4 to 65.2] | 54.4 [43.6 to 65.0] | 61.3 [50.6 to 71.2] | 67.0 [56.2 to 76.7] | 49.5 [39.1 to 59.9] | 61.5 [53.4 to 69.2] | 37.0 [19.4 to 57.6] | 79.1 [64.0 to 90.0] | 42.4 [25.5 to 60.8] | 57.9 [44.1 to 70.9] | 50.0 [35.5 to 64.5]

3. Secondary Outcome: Average Percentage of Subjects Achieving a TNA Response of a Predefined Threshold Value Between Days 63 and 100 (Inclusive).
Description: as for outcome 1
Time Frame: Days 63 to 100
Population: Participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- BioThrax - Days 63-100 Immunogenicity: Participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Male: Male participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Female: Female participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - ≤ 30 Years of Age: Participants ≤ 30 Years of Age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - > 30 Years of Age: Participants > 30 Years of Age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Caucasian: Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Non-Caucasian: Non-Caucasian participants 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Site 01: Participants enrolled at Site 01, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Site 02: Participants enrolled at Site 02, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Site 03: Participants enrolled at Site 03, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
- BioThrax - Site 04: Participants enrolled at Site 04, 18 to 65 years of age who received all three doses of BioThrax (0.5 mL) subcutaneously (SC) within the allowable time window (±2 days for Days 14 and 28) and had a blood sample collected for immunogenicity testing on Day 63 ± 2 days, Day 70 ± 2 days, Day 84 ± 3 days, and Day 100 ± 3 days, inclusive. Subjects with key protocol deviations that may have impacted assessment of immune response or sample testing (as determined by the Sponsor) on Days 63, 70, 84, or 100 were excluded.
Arm/Group | BioThrax - Days 63-100 Immunogenicity | BioThrax - Male | BioThrax - Female | BioThrax - ≤ 30 Years of Age | BioThrax - > 30 Years of Age | BioThrax - Caucasian | BioThrax - Non-Caucasian | BioThrax - Site 01 | BioThrax - Site 02 | BioThrax - Site 03 | BioThrax - Site 04
Number analyzed (Participants) | 165 | 82 | 83 | 77 | 88 | 141 | 24 | 36 | 30 | 52 | 47
percentage of participants | 52.7 [44.8 to 60.5] | 50.0 [38.7 to 61.3] | 55.4 [44.1 to 66.3] | 58.4 [46.6 to 69.6] | 47.7 [37.0 to 58.6] | 56.0 [47.4 to 64.4] | 33.3 [15.6 to 55.3] | 75.0 [57.8 to 87.9] | 36.7 [19.9 to 56.1] | 51.9 [37.6 to 66.0] | 46.8 [32.1 to 61.9]

4. Secondary Outcome: Incidence of Injection Site Reactions by Severity (Mild, Moderate, Severe) From Subject Diary Cards
Description: Injection site reactions (warmth, tenderness, itching, pain, arm motion limitation, redness, lump, swelling, and bruise) were evaluated by using a web-enabled subject diary. Subjects assessed the severity of warmth, tenderness, itching, pain, arm motion limitation, lump, and bruise as absent, mild, moderate, or severe based on the degree of interference with daily activities. Severity of redness and swelling were based on the diameter of the affected area. Severe injection site reactions were recorded as adverse events by the investigator site staff after confirmation with the subject.
Time Frame: Web-enabled diaries were completed for 7 days after each of three injections (Days 0, 14, and 28).
Population: The reporting group was subjects who had any diary data available during the 7-day-post-vaccination period (i.e., n=196, n=196, and n=193, for the1st, 2nd, and 3rd post-vaccination periods, respectively).
Measure: Number; unit: participants
Groups:
- BioThrax 1st Vaccination - No Reaction; BioThrax 1st Vaccination - Mild Reaction; BioThrax 1st Vaccination - Moderate Reaction; BioThrax 1st Vaccination - Severe Reaction; BioThrax 1st Vaccination - Total of Reactions; BioThrax 2nd Vaccination - No Reaction; BioThrax 2nd Vaccination - Mild Reaction; BioThrax 2nd Vaccination - Moderate Reaction; BioThrax 2nd Vaccination - Severe Reaction; BioThrax 2nd Vaccination - Total of Reactions; BioThrax 3rd Vaccination - No Reaction; BioThrax 3rd Vaccination - Mild Reaction; BioThrax 3rd Vaccination - Moderate Reaction; BioThrax 3rd Vaccination - Severe Reaction; BioThrax 3rd Vaccination - Total of Reactions: The incidence of injection site reactions was evaluated in the population of subjects who had any diary data available during the 7-day-post-vaccination period
Arm/Group | BioThrax 1st Vaccination - No Reaction | BioThrax 1st Vaccination - Mild Reaction | BioThrax 1st Vaccination - Moderate Reaction | BioThrax 1st Vaccination - Severe Reaction | BioThrax 1st Vaccination - Total of Reactions | BioThrax 2nd Vaccination - No Reaction | BioThrax 2nd Vaccination - Mild Reaction | BioThrax 2nd Vaccination - Moderate Reaction | BioThrax 2nd Vaccination - Severe Reaction | BioThrax 2nd Vaccination - Total of Reactions | BioThrax 3rd Vaccination - No Reaction | BioThrax 3rd Vaccination - Mild Reaction | BioThrax 3rd Vaccination - Moderate Reaction | BioThrax 3rd Vaccination - Severe Reaction | BioThrax 3rd Vaccination - Total of Reactions
Number analyzed (Participants) | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 193 | 193 | 193 | 193 | 193
participants
  Warmth | 93 | 94 | 9 | 0 | 103 | 85 | 96 | 14 | 1 | 111 | 101 | 88 | 4 | 0 | 92
  Tenderness | 11 | 134 | 49 | 2 | 185 | 11 | 126 | 57 | 2 | 185 | 36 | 139 | 18 | 0 | 157
  Itching | 167 | 27 | 1 | 1 | 29 | 118 | 65 | 12 | 1 | 78 | 121 | 65 | 7 | 0 | 72
  Pain | 26 | 123 | 45 | 2 | 170 | 34 | 110 | 50 | 2 | 162 | 80 | 100 | 13 | 0 | 113
  Arm Motion Limitation | 102 | 68 | 22 | 4 | 94 | 102 | 66 | 27 | 1 | 94 | 137 | 51 | 5 | 0 | 56
  Redness | 115 | 68 | 12 | 1 | 81 | 84 | 80 | 30 | 2 | 112 | 109 | 70 | 14 | 0 | 84
  Swelling | 111 | 78 | 7 | 0 | 85 | 90 | 85 | 21 | 0 | 106 | 111 | 73 | 9 | 0 | 82
  Lump | 82 | 102 | 11 | 1 | 114 | 62 | 109 | 23 | 2 | 134 | 76 | 107 | 10 | 0 | 117
  Bruise | 173 | 23 | 0 | 0 | 23 | 162 | 31 | 2 | 1 | 34 | 171 | 21 | 1 | 0 | 22

5. Secondary Outcome: Percentage of Injection Site Reactions by Severity (Mild, Moderate, Severe) From Subject Diary Cards
Description: as for outcome 4
Time Frame: Web-enabled diaries were completed for 7 days after each of three injections (Days 0, 14, and 28).
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | BioThrax 1st Vaccination - No Reaction | BioThrax 1st Vaccination - Mild Reaction | BioThrax 1st Vaccination - Moderate Reaction | BioThrax 1st Vaccination - Severe Reaction | BioThrax 1st Vaccination - Total of Reactions | BioThrax 2nd Vaccination - No Reaction | BioThrax 2nd Vaccination - Mild Reaction | BioThrax 2nd Vaccination - Moderate Reaction | BioThrax 2nd Vaccination - Severe Reaction | BioThrax 2nd Vaccination - Total of Reactions | BioThrax 3rd Vaccination - No Reaction | BioThrax 3rd Vaccination - Mild Reaction | BioThrax 3rd Vaccination - Moderate Reaction | BioThrax 3rd Vaccination - Severe Reaction | BioThrax 3rd Vaccination - Total of Reactions
Number analyzed (Participants) | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 193 | 193 | 193 | 193 | 193
percentage of participants
  Warmth | 47.4 | 48.0 | 4.6 | 0 | 52.6 | 43.4 | 49.0 | 7.1 | 0.5 | 56.6 | 52.3 | 45.6 | 2.1 | 0 | 47.7
  Tenderness | 5.6 | 68.4 | 25.0 | 1.0 | 94.4 | 5.6 | 64.3 | 29.1 | 1.0 | 94.4 | 18.7 | 72.0 | 9.3 | 0 | 81.3
  Itching | 85.2 | 13.8 | 0.5 | 0.5 | 14.8 | 60.2 | 33.2 | 6.1 | 0.5 | 39.8 | 62.7 | 33.7 | 3.6 | 0 | 37.3
  Pain | 13.3 | 62.8 | 23.0 | 1.0 | 86.7 | 17.3 | 56.1 | 25.5 | 1.0 | 82.7 | 41.5 | 51.8 | 6.7 | 0 | 58.5
  Arm Motion Limitation | 52.0 | 34.7 | 11.2 | 2.0 | 48.0 | 52.0 | 33.7 | 13.8 | 0.5 | 48.0 | 71.0 | 26.4 | 2.6 | 0 | 29.0
  Redness | 58.7 | 34.7 | 6.1 | 0.5 | 41.3 | 42.9 | 40.8 | 15.3 | 1.0 | 57.1 | 65.5 | 36.3 | 7.3 | 0 | 43.5
  Swelling | 56.6 | 39.8 | 3.6 | 0 | 43.4 | 45.9 | 43.4 | 10.7 | 0 | 54.1 | 57.5 | 37.8 | 4.7 | 0 | 42.5
  Lump | 41.8 | 52.0 | 5.6 | 0.5 | 58.2 | 31.6 | 55.6 | 11.7 | 1.0 | 68.4 | 39.4 | 55.4 | 5.2 | 0 | 60.6
  Bruise | 88.3 | 11.7 | 0 | 0 | 11.7 | 82.7 | 15.8 | 1.0 | 0.5 | 17.3 | 88.6 | 10.9 | 0.5 | 0 | 11.4

6. Secondary Outcome: Incidence of Systemic Reactions by Severity (Mild, Moderate, Severe) From Subject Diary Cards
Description: Systemic reactions (fatigue/ tiredness, muscle ache, headache, and fever) were evaluated by using a web-enabled subject diary. Subjects assessed severity as absent, mild, moderate, or severe based on the degree of interference with daily activities. Severity of fever was assessed using a grading scale. Severe systemic reactions were to be recorded as adverse events by the investigator site staff after confirmation with the subject.
Time Frame: Web-enabled diaries were completed for 7 days after each of three injections (Days 0, 14, and 28).
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- BioThrax 1st Vaccination - No Reaction; BioThrax 1st Vaccination - Mild Reaction; BioThrax 1st Vaccination - Moderate Reaction; BioThrax 1st Vaccination - Severe Reaction; BioThrax 1st Vaccination - Total of Reactions; BioThrax 2nd Vaccination - No Reaction; BioThrax 2nd Vaccination - Mild Reaction; BioThrax 2nd Vaccination - Moderate Reaction; BioThrax 2nd Vaccination - Severe Reaction; BioThrax 2nd Vaccination - Total of Reactions; BioThrax 3rd Vaccination - No Reaction; BioThrax 3rd Vaccination - Mild Reaction; BioThrax 3rd Vaccination - Moderate Reaction; BioThrax 3rd Vaccination - Severe Reaction; BioThrax 3rd Vaccination - Total of Reactions: The incidence of systemic reactions was evaluated in the population of subjects who had any diary data available during the 7-day-post-vaccination period
Arm/Group | BioThrax 1st Vaccination - No Reaction | BioThrax 1st Vaccination - Mild Reaction | BioThrax 1st Vaccination - Moderate Reaction | BioThrax 1st Vaccination - Severe Reaction | BioThrax 1st Vaccination - Total of Reactions | BioThrax 2nd Vaccination - No Reaction | BioThrax 2nd Vaccination - Mild Reaction | BioThrax 2nd Vaccination - Moderate Reaction | BioThrax 2nd Vaccination - Severe Reaction | BioThrax 2nd Vaccination - Total of Reactions | BioThrax 3rd Vaccination - No Reaction | BioThrax 3rd Vaccination - Mild Reaction | BioThrax 3rd Vaccination - Moderate Reaction | BioThrax 3rd Vaccination - Severe Reaction | BioThrax 3rd Vaccination - Total of Reactions
Number analyzed (Participants) | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 193 | 193 | 193 | 193 | 193
participants
  Fatigue/Tiredness | 138 | 48 | 10 | 0 | 58 | 135 | 48 | 12 | 1 | 61 | 151 | 38 | 4 | 0 | 42
  Muscle Ache | 86 | 90 | 19 | 1 | 110 | 101 | 67 | 27 | 1 | 95 | 125 | 63 | 5 | 0 | 68
  Headache | 147 | 38 | 9 | 2 | 49 | 140 | 40 | 15 | 1 | 56 | 143 | 38 | 12 | 0 | 50
  Fever | 195 | 0 | 1 | 0 | 1 | 196 | 0 | 0 | 0 | 0 | 192 | 1 | 0 | 0 | 1

7. Secondary Outcome: Percentage of Systemic Reactions by Severity (Mild, Moderate, Severe) From Subject Diary Cards
Description: as for outcome 6
Time Frame: Web-enabled diaries were completed for 7 days after each of three injections (Days 0, 14, and 28).
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | BioThrax 1st Vaccination - No Reaction | BioThrax 1st Vaccination - Mild Reaction | BioThrax 1st Vaccination - Moderate Reaction | BioThrax 1st Vaccination - Severe Reaction | BioThrax 1st Vaccination - Total of Reactions | BioThrax 2nd Vaccination - No Reaction | BioThrax 2nd Vaccination - Mild Reaction | BioThrax 2nd Vaccination - Moderate Reaction | BioThrax 2nd Vaccination - Severe Reaction | BioThrax 2nd Vaccination - Total of Reactions | BioThrax 3rd Vaccination - No Reaction | BioThrax 3rd Vaccination - Mild Reaction | BioThrax 3rd Vaccination - Moderate Reaction | BioThrax 3rd Vaccination - Severe Reaction | BioThrax 3rd Vaccination - Total of Reactions
Number analyzed (Participants) | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 196 | 193 | 193 | 193 | 193 | 193
percentage of participants
  Fatigue/Tiredness | 70.4 | 24.5 | 5.1 | 0 | 29.6 | 68.9 | 24.5 | 6.1 | 0.5 | 31.1 | 78.2 | 19.7 | 2.1 | 0 | 21.8
  Muscle Ache | 43.9 | 45.9 | 9.7 | 0.5 | 56.1 | 51.5 | 34.2 | 13.8 | 0.5 | 48.5 | 64.8 | 32.6 | 2.6 | 0 | 35.2
  Headache | 75.0 | 19.4 | 4.6 | 1.0 | 25.0 | 71.4 | 20.4 | 7.7 | 0.5 | 28.6 | 74.1 | 19.7 | 6.2 | 0 | 25.9
  Fever | 99.25 | 0 | 0.5 | 0 | 0.5 | 100 | 0 | 0 | 0 | 0 | 99.5 | 0.5 | 0 | 0 | 0.5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of screening up to 100 days post dose.
Groups:
- ITT Population: Participants 18 to 65 years of age who received at least one dose of BioThrax (0.5 mL) subcutaneously (SC).
Arm/Group | ITT Population
Serious Adverse Events (participants affected / at risk) | 2/200
Other Adverse Events (participants affected / at risk) | 109/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=200)
Obesity (Metabolism and nutrition disorders) | 1 (1) — The participant was hospitalized due to elective gastric bypass for morbid obesity. The event was assessed by the principal investigator as not related to vaccination. The event resolved without sequelae, and the subject completed the study.
Aura (Nervous system disorders) | 1 (1) — The participant experienced a visual aura without headache. The event was assessed by the principal investigator as not related to vaccination. The event resolved without sequelae, and the subject completed the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=200)
Upper respiratory tract infection (Infections and infestations) | 37 (44)
Headache (Nervous system disorders) | 25 (31)
Fatigue (General disorders) | 13 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (14)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Nasopharyngitis (Infections and infestations) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor is responsible for public disclosure of study data. Any proposed publication is subject to review agreed between Biomedical Advanced Research and Development Authority (BARDA)and Emergent; between Emergent and the contract research organizations (CROs)/vendors; and between the CROs and the site Principal Investigator. Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.